CLINICAL TRIAL: NCT03221933
Title: Phase Ⅱ Clinical Study of Recombinant Human Growth Hormone Injection（JINTOPIN AQ）for Short Children With Small for Gestational Age(SGA)
Brief Title: A Study of Recombinant Human Growth Hormone Injection（JINTOPIN AQ）for Short Children With Small for SGA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Tongji Hospital (Other); Beijing Children's Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Shanghai Children's Hospital (Other); The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GenSci 030 CT-II
Record Dates: First submitted 2017-07-16; First posted 2017-07-19 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-07

CONDITIONS: Small for Gestational Age Infant
MeSH Terms: interventions — Human Growth Hormone; Population Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Somatropin Injection low dose group (Experimental): 0.23mg/kg /wk，inject for seven divided doses.
  Interventions: Biological: Somatropin Injection low dose group; Biological: Somatropin Injection high dose group
- Somatropin Injection high dose group (Experimental): 0.46mg/kg /wk，inject for seven divided doses.
  Interventions: Biological: Somatropin Injection low dose group; Biological: Somatropin Injection high dose group

INTERVENTIONS:
Biological: Somatropin Injection low dose group — 0.23mg/kg /wk，inject for seven divided doses
Biological: Somatropin Injection high dose group — 0.46mg/kg /wk，inject for seven divided dose

SUMMARY:
To preliminary assess the efficacy and safety of recombinant human growth hormone injection on the treatment of small for gestational age (SGA), and determine the best dose.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of small for gestational age, SGA.
* Chronological age between 2-6.5 years in girls and 2-7.5 years in boys. Both genders.
* Prepubertal stage (Tanner I).
* Without catch-up growth in two years after birth.
* Height was lower than the mean -2SD of the values of normal children of the same age and gender when participating in the study.
* A GH peak concentration >10µg/L in a provocative test within a year before participate in the study.
* Bone age<Chronological age+1.
* Normal glucose regulation：Fasting blood-glucose < 5.6mmol/L and 2-hour postprandial blood glucose< 7.8mmol/L.
* Gestational age≥Gestational age≥ 36weeks + 4days.
* Never accepted growth hormone treatment.
* The subjects and their guardians signed informed consent.

Exclusion Criteria:

* Subjects with Liver and renal insufficiency (ALT > 2 times of upper limit of normal value, Cr> upper limit of normal value).
* Patients with positive for antibodies to hepatitis B core (anti-HBc), hepatitis B surface antigen (HBsAg) or hepatitis B e antigen (HBeAg)。
* Known highly allergic constitution or allergic to the test drug.
* Subjects with diabetes, severe cardiopulmonary and pulmonary disease, and hematological diseases, malignant tumors, or systemic infection, immunocompromised patients and patients with psychosis.
* Subjects with other types of abnormal growth and development, such as Turner syndrome, constitutional delay of puberty, Laron syndrome, growth hormone receptor deficiency.
* Subjects who have received the treatment of Somatropin or took part in other clinical trial study within 3 months.
* Other conditions which in the opinion of the investigator preclude enrollment into the study.

Ages: 24 Months to 90 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Height standard deviation score for chronological age (Ht SDSCA) | 26 weeks
  HtSDSCA = (height-reference mean for CA) / reference SD for CA (refers to the height value at particular timepoint)
Height standard deviation score for chronological age (Ht SDSCA) | 52 weeks
  HtSDSCA = (height-reference mean for CA) / reference SD for CA (refers to the height value at particular timepoint)
Height standard deviation score for chronological age (Ht SDSCA) | 78 weeks
  HtSDSCA = (height-reference mean for CA) / reference SD for CA (refers to the height value at particular timepoint)
Height standard deviation score for chronological age (Ht SDSCA) | 104 weeks
  HtSDSCA = (height-reference mean for CA) / reference SD for CA (refers to the height value at particular timepoint)

SECONDARY OUTCOMES:
ΔHtSDSCA | 26 weeks， 52 weeks，78 weeks and 104 weeks
  Change in height SDS for chronological age (Ht SDSCA)
Change in HV | 26 weeks， 52 weeks，78 weeks and 104 weeks
  Change in annualized height velocity (HV)
Change in bone age maturation | 26 weeks， 52 weeks，78 weeks and 104 weeks
Change in mole ratio of IGF-1 and IGFBP-3 | 26 weeks， 52 weeks，78 weeks and 104 weeks
Change in PAH | 26 weeks， 52 weeks，78 weeks and 104 weeks
  Change in prediction of adult height (PAH)
Change in obesity prevalence | 26 weeks， 52 weeks，78 weeks and 104 weeks
Change in overweight | 26 weeks， 52 weeks，78 weeks and 104 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Luo, Principal Investigator — Department of Pediatrics of Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology
Locations (5):
- China (5):
  - Tongji Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - The first affiliated Hospital with Nanjing Medical Universit, Nanjing, Jiangsu
  - Children's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Beijing Children's Hospital of Capital Medical University, Beijing
  - Shanghai Children's Hospital, Shanghai